CLINICAL TRIAL: NCT06470256
Title: Palliative Hepatectomy Combined With Targeted Therapy and Immunotherapy for Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhiyong Huang (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Zhongnan Hospital (Other); Renmin Hospital of Wuhan University (Other); Taihe Hospital (Other); Hubei Cancer Hospital (Other); Xiangyang Central Hospital (Other); Wuhan Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhiyong Huang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: aHCC-PHTI-TJ01
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: HCC; Palliative Hepatectomy; Immunotherapy; Targeted therapy
MeSH Terms: interventions — durvalumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palliative Hepatectomy Combined With Targeted Therapy and Immunotherapy (Experimental): Reduce tumor burden by over 90% through palliative hepatectomy . Starting two weeks post-surgery, patients began intravenous infusions of the PD-L1 monoclonal antibody, Durvalumab, at a dosage of 1500 mg every three weeks. Three weeks post-surgery, patients commenced oral administration of the targeted therapy, Lenvatinib, with a dosage based on body weight: 8 mg (≤60 kg) or 12 mg (>60 kg), once daily. The use of Durvalumab and Lenvatinib continued until the primary endpoint or other criteria specified in the protocol for terminating the study treatment.
  Interventions: Procedure: Palliative Hepatectomy; Drug: Durvalumab; Drug: Lenvatinib

INTERVENTIONS:
Procedure: Palliative Hepatectomy — Patients will receive TACE, HAIC, or 90Y-SIRT combined with Lenvatinib and Durvalumab. After receiving three months of combined treatment, patients in the SD or PD stage who have poor efficacy evaluated by imaging will undergo palliative hepatectomy.
  Palliative Hepatectomy:① Intrahepatic metastasis: complete lesion resection of the main tumor on one side of the liver; ② Extrahepatic metastasis: complete lesion resection of intrahepatic lesions; ③ Merge portal vein tumor thrombus or hepatic vein tumor thrombus: remove the tumor thrombus and completely remove the intrahepatic lesions. And reduce the tumor burden by more than 90% through surgical resection.
Drug: Durvalumab — Starting two weeks post-surgery, patients began intravenous infusions of the PD-L1 monoclonal antibody, Durvalumab.
  Other Names: IMFINZ
Drug: Lenvatinib — Three weeks post-surgery, patients commenced oral administration of Lenvatinib.
  Other Names: LENVIMA

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the most common malignant tumors and the leading cause of cancer-related death worldwide. Surgical resection has always been the best hope for long-term survival of patients with HCC. However, due to the fact that most patients are already in the middle and late stages of treatment, only about 20% of patients have the opportunity to undergo surgical resection. Palliative cytoreductive surgery has been used in the treatment of a variety of malignant tumors, but it is not recommended for the treatment of HCC. Under the premise of targeted therapy and immunotherapy, palliative hepatectomy can reduce tumor burden and may further improve the therapeutic effect of HCC. The aim of this study is to explore whether palliative hepatectomy combined with targeted therapy and immunotherapy can improve the therapeutic effect of advanced HCC, ultimately prolong the survival time of patients, and provide a new treatment direction for patients with advanced HCC.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, single-arm clinical study aimed at evaluating targeted therapy and immunotherapy combined with palliative hepatectomy for the treatment of advanced hepatocellular carcinoma. Patients who have been assessed as stage B or C of Barcelona Clinic Liver Cancer (BCLC) will receive local treatment (transcatheter arterial chemoembolization (TACE) or transcatheter arterial chemoembolization (HAIC)) or 90Y-SIRT (yttrium-90 selective internal radiation therapy) combined with Lenvatinib and Durvalumab. After receiving three months of combined treatment, patients in the stable disease (SD) or progressive disease (PD) stage who have poor efficacy evaluated by imaging will undergo palliative hepatectomy; patients in the complete response (CR) or partial response (PR) stage after imaging evaluation will be excluded and continue to receive systematic treatment. Patients need to discontinue targeted therapy and immunotherapy one week before surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 75 years (inclusive).
2. No prior systemic antitumor treatment or surgical treatment.
3. Clinical or pathological diagnosis of hepatocellular carcinoma (HCC).
4. The primary liver lesion is mainly isolated liver tumors, with a tumor burden exceeding 90% of the total tumor burden, and technically capable of complete resection. Simultaneously merging ① intrahepatic metastasis: the number of metastatic tumors is ≥ 3 and the sum of tumor diameters is ≤ 3cm; Or ② Extrahepatic metastasis: Extrahepatic metastasis does not exceed one organ, metastatic tumors do not exceed three, and the total diameter does not exceed 3cm. Or ③ if combined with portal vein tumor thrombus or hepatic vein tumor thrombus, it can be removed or completely removed together with the main tumor, and the tumor thrombus does not enter the superior mesenteric vein or inferior vena cava.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1, without significant organ dysfunction.
6. Child-Pugh class A.
7. HBV-DNA less than 1*10^5 copies/ml and undergoing antiviral therapy.
8. Important organ functions meeting the following criteria: White Blood Cell (WBC) ≥2.5 × 10^9/L ;Platelet (PLT) ≥75 × 10^9/L;Hemoglobin (HB) ≥ 9g/dL;Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤ 3*ULN, Total Bilirubin ≤ 3*ULN; International Normalized Ratio (INR) ≤ 1.5*ULN; Prothrombin Time ≤ 1.5*ULN; Creatinine ≤ 1.5*ULN.
9. Expected survival time of more than 3 months.
10. According to the RECIST v1.1 standard, postoperative patients with at least one longest diameter of 1 cm or more measurable tumors.
11. Willing to provide informed consent.

Exclusion Criteria:

1. History of or concurrent active malignancy (excluding malignancies that have been cured for over 5 years or in situ cancers that can be completely cured with adequate treatment).
2. Presence of central nervous system metastasis or a history of brain metastasis.
3. History of organ transplantation.
4. History of surgery in the head, chest, or abdomen within the past six months.
5. Child-Pugh class C liver function or massive ascites.
6. Ongoing active infection within 7 days after completion of systemic antibiotic therapy.
7. Active coronary artery disease, severe/unstable angina, or newly diagnosed angina or myocardial infarction within the past 12 months before enrollment.
8. Thrombotic or embolic events within the past 12 months, such as cerebrovascular accidents (including transient ischemic attacks), pulmonary embolism, or deep vein thrombosis.
9. New York Heart Association (NYHA) class II or above congestive heart failure.
10. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), positive syphilis serology, untreated active hepatitis (defined as HBV-DNA ≥ 10^5 copies/ml; HCV-RNA higher than the lower limit of detection for the assay).
11. Any active, known, or suspected autoimmune disease. Stable subjects not requiring systemic immunosuppressive therapy may be included, such as those with type 1 diabetes, hypothyroidism requiring only hormone replacement therapy, and skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis, and alopecia).
12. Interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, and acute pneumonia).
13. Pregnant or lactating women or females with a positive pregnancy test prior to the first dose who have the potential for pregnancy.
14. The investigator deems the subject inappropriate for participation in this clinical study due to any clinical or laboratory abnormalities or compliance issues.
15. Severe psychological or mental abnormalities.
16. Participation in another drug clinical trial within the past 4 weeks.
17. Other reasons that the investigator considers unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6 weeks after first dose of Durvalumab
  ORR refers to the proportion of patients whose tumors shrink to a certain amount and maintain for a certain period of time (6 weeks after first dose of Durvalumab), including CR+PR cases. CR (complete response): disappearance of all target lesions, PR (partial response): reduction of the sum of the length and diameter of the baseline lesions by ≥30%.

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 2 year
  OS was defined as time from diagnosis to death from any cause or the last follow-up
Progression Free Survival (PFS) | 18 months
  PFS refers to the time from subject enrollment to disease progression according the Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1) or death

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Huang, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China